CLINICAL TRIAL: NCT03861728
Title: Avenova for the Treatment of Viral Conjunctivitis
Brief Title: Viral Conjunctivitis Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Pandemic
Sponsor: University of Miami (Other)
Collaborators: NovaBay Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Wendy Lee, Associate Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 20170064
Record Dates: First submitted 2018-12-11; First posted 2019-03-04 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Viral Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Viral

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: A second investigator will randomize the patient to Treatment vs Placebo on initial visit. This "second investigator" will not be involved in screening or follow-up patient visits. At the end of the study the patient arms will be unmasked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Viral Conjunctivitis Treatment (Experimental): Patients with viral conjunctivitis as defined by a + AdenoPlus test and clinical symptoms and signs of viral conjunctivitis who will be treated with 0.01% Hypochlorous acid
  Interventions: Device: 0.01% Hypochlorous acid
- Viral Conjunctivitis Placebo (Placebo Comparator): Patients with viral conjunctivitis as defined by a + AdenoPlus test and clinical symptoms and signs of viral conjunctivitis who will be treated with Basic Sterile Saline
  Interventions: Other: Placebo

INTERVENTIONS:
Device: 0.01% Hypochlorous acid — Randomized to treatment 0.01% Hypochlorous acid four times a day to the affected eye for 2 weeks. (Avenova is a FDA approved device)
  Other Names: Avenova
  Arms: Viral Conjunctivitis Treatment
Other: Placebo — Placebo to be used four times a day to the affected eye for 2 weeks
  Other Names: Basic Sterile Saline
  Arms: Viral Conjunctivitis Placebo

SUMMARY:
The objective of this study is to determine the efficacy Avenova® (0.01% hypochlorous acid) in the treatment of viral conjunctivitis. The investigators hypothesize that patients treated with Avenova® will have a quicker resolution of their ocular signs and symptoms of Viral Conjunctivitis compared with artificial tears.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the Bascom Palmer Eye Institute
* Clinical diagnosis of viral conjunctivitis
* Symptoms less than 1 week duration

Exclusion Criteria:

* history of allergic conjunctivitis
* history of herpetic eye disease
* concurrent diagnosis of bacterial conjunctivitis (based off microbiology plating)
* Immunocompromised / Immunosuppressed patients
* Patients with HIV
* pregnant women
* prisoners
* adults who are unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-02-08 (Actual); Study Completion 2020-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Lee, MD, Principal Investigator — Bascom Palmer Eye Institute, University of Miami
Locations (1):
- University of Miami Bascom Palmer Eye Institute, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Debabov D, Noorbakhsh C, Wang L, et al. Avenova™ with Neutrox™ (pure 0.01% HOCl) compared with OTC product (0.02% HOCl). NovaBay Pharmaceuticals, Inc., Emeryville, California, USA
- [Result] Kim HJ, Lee JG, Kang JW, Cho HJ, Kim HS, Byeon HK, Yoon JH. Effects of a low concentration hypochlorous Acid nasal irrigation solution on bacteria, fungi, and virus. Laryngoscope. 2008 Oct;118(10):1862-7. doi: 10.1097/MLG.0b013e31817f4d34. PMID 18677274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Viral Conjunctivitis Treatment | Viral Conjunctivitis Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of treatment or placebo and returned for follow up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Viral Conjunctivitis Treatment | Viral Conjunctivitis Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Median (Full Range); unit: years] | 40 [22 to 74] | 48 [22 to 56] | 40 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Duration of Symptoms Prior to Presentation [Median (Full Range); unit: days] | 3 [1 to 5] | 1 [1 to 5] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Resolution of Viral Conjunctivitis
Description: This is the number of participants who on day 7 (+/-1 days) had on clinical examination a 0 or 1 on the follicular conjunctivitis scale and 0 or 1 on the conjunctival injection scale.
Time Frame: Up to 8 days
Population: All participants who received at least one dose of treatment or placebo and returned for follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Conjunctivitis Treatment | Viral Conjunctivitis Placebo
Number analyzed (Participants) | 6 | 5
Participants | 3 | 3

2. Secondary Outcome: Number of Participants With Symptomatic Resolution of Viral Conjunctivitis
Description: This is the number of participants who on day 7 (+/-1 days) answered on clinical questionaire "none" or "mild" to each of the following list of 7 symptoms: "overall symptoms that affect your daily activities", "itching", "tearing", "pain", "feeling that your lids are stuck together in the morning", "sensitivity to light", "blurry vision"
Time Frame: Up to 8 days
Population: All participants who received at least one dose of treatment or placebo and returned for follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Conjunctivitis Treatment | Viral Conjunctivitis Placebo
Number analyzed (Participants) | 6 | 5
Participants | 2 | 4

3. Secondary Outcome: Number of Participants With Undetectable Adenoviral DNA
Description: This is the number of participants who on day 7 (+/-1 days) had undetectable adenoviral DNA by quantitative Polymerase Chain Reaction (qPCR) (Ct > 35)
Time Frame: Up to 8 days
Population: All participants who received at least one dose of treatment or placebo and returned for follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Viral Conjunctivitis Treatment | Viral Conjunctivitis Placebo
Number analyzed (Participants) | 6 | 5
Participants | 3 | 1

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Viral Conjunctivitis Treatment | Viral Conjunctivitis Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 0/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Viral Conjunctivitis Treatment (N=6) | Viral Conjunctivitis Placebo (N=5)
HSV Keratitis (Eye disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination led to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT03861728/Prot_SAP_001.pdf